CLINICAL TRIAL: NCT06235619
Title: CT Anatomical Characteristics of the Aortic Arch in Subjects With or Without Aneurysms Requiring Treatment
Brief Title: Arch Size Study for Anatomical Variations
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Germano Melissano, Prof., IRCCS San Raffaele
Other Study IDs: archsize
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Aortic Arch; Aneurysm; Dissection, Aortic
Keywords: Aortic arch; Bovine arch; Thoracic aortic disease
MeSH Terms: conditions — Aneurysm; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non aneurysm patients: CT anatomical characteristics of the aortic arch in subjects without aneurysms requiring treatment.
- Aneurysm patients: CT anatomical characteristics of the aortic arch in subjects withaneurysms requiring treatment.

SUMMARY:
The aortic arch with a common origin of the innominate and left carotid artery (CILCA) prevalence in the general population is 13.6%. Its reputation as a benign anatomical variant has been ultimately shattered by further studies that identified the CILCA arch as a potential marker for thoracic aortic disease (TAD) The aim of this work is to report the CT anatomical characteristics of the aortic arch in subjects with or without aneurysms requiring treatment, in 5 major European cardiovascular centers.

ELIGIBILITY:
Inclusion Criteria:

all patients with aortic arch CT scan at investigating centers

Exclusion Criteria:

none

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of the study is the general population undergoing Angio CT scan both the thoracic aorta
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
difference from baseline of aortic arch anomalies | 30 day
  record of anatomical variations of the aortic arch

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided